CLINICAL TRIAL: NCT00371007
Title: MK0431 Early Phase II Double-blind Study - Type 2 Diabetes Mellitus
Brief Title: MK-0431 Early Phase II Double-blind Study - Type 2 Diabetes Mellitus (0431-043)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-043; 2006_028
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0431, sitagliptin phosphate / Duration of Treatment: 12 Weeks
Drug: Comparator : placebo (unspecified) / Duration of Treatment: 12 Weeks

SUMMARY:
A clinical study to determine the safety and efficacy of MK-0431 in patients with Type 2 diabetes mellitus who have inadequate glycemic control on diet/exercise therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients have type 2 diabetes mellitus
* On diet/exercise therapy

Exclusion Criteria:

* Patients have type 1 diabetes mellitus

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126
Dates: Start 2004-06-01 (Actual); Primary Completion 2005-04-25 (Actual); Study Completion 2005-04-25 (Actual)

PRIMARY OUTCOMES:
HbA1c, safety and tolerability

SECONDARY OUTCOMES:
Plasma glucose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Nonaka K, Kakikawa T, Sato A, Okuyama K, Fujimoto G, Kato N, Suzuki H, Hirayama Y, Ahmed T, Davies MJ, Stein PP. Efficacy and safety of sitagliptin monotherapy in Japanese patients with type 2 diabetes. Diabetes Res Clin Pract. 2008 Feb;79(2):291-8. doi: 10.1016/j.diabres.2007.08.021. Epub 2007 Oct 22. PMID 17933414
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html